CLINICAL TRIAL: NCT05543642
Title: The COvid19 VaccinE Response and Co-Administration in Rheumatology Patients (COVER-CoAd)
Brief Title: The COVID-19 VaccinE Response and Co-Administration in Rheumatology Patients (COVER-CoAd)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kevin Winthrop, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: COVER-CoAd
Record Dates: First submitted 2022-09-02; First posted 2022-09-16 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Rheumatic Diseases
MeSH Terms: conditions — Rheumatic Diseases | interventions — Hepatitis A Vaccines; Boostrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1 (control group, sequential administration) (Active Comparator): Individuals with other chronic conditions and not active rheumatic disease (defined as being treated), who are eligible to receive their tdap booster and hepA vaccines, and receiving a COVID-19 booster vaccination.
  This arm will receive sequential administration of both tdap booster and hepA vaccinations.
  Interventions: Biological: Hepatitis A vaccine; Biological: Diphtheria, pertussis, and tetanus booster vaccine
- Arm 2 (co-administration group) (Active Comparator): Individuals with other chronic conditions and not active rheumatic disease (defined as being treated), who are eligible to receive their tdap booster and hepA vaccines, and receiving a COVID-19 booster vaccination.
  This arm will receive co-administration of hepA vaccination.
  Interventions: Biological: Hepatitis A vaccine
- Arm 3 (co-administration group) (Active Comparator): Individuals with other chronic conditions and not active rheumatic disease (defined as being treated), who are eligible to receive their tdap booster and hepA vaccines, and receiving a COVID-19 booster vaccination.
  This arm will receive co-administration of tdap booster vaccination.
  Interventions: Biological: Diphtheria, pertussis, and tetanus booster vaccine
- Arm 4 (Inflammatory arthritis patients using DMARDS) (No Intervention): Individuals with inflammatory arthritis patients using DMARDS, who are eligible to receive their tdap booster and hepA vaccines, and receiving a COVID-19 booster vaccination.
  This arm will only receive the standard of care COVID-19 booster vaccination.

INTERVENTIONS:
Biological: Hepatitis A vaccine — Vaccination series administered to prevent hepA infection.
  Other Names: Havrix
  Arms: Arm 1 (control group, sequential administration); Arm 2 (co-administration group)
Biological: Diphtheria, pertussis, and tetanus booster vaccine — Vaccination booster administered to prevent diphtheria, pertussis, and tetanus
  Other Names: Boostrix
  Arms: Arm 1 (control group, sequential administration); Arm 3 (co-administration group)

SUMMARY:
Based on the experience with influenza, pneumococcal, and shingles vaccinations in rheumatic disease populations, it is clear that some disease modifying anti-rheumatic drugs and the immunomodulatory therapies used to treat immune-mediated inflammatory diseases have the capacity to blunt immune responses to COVID-19 vaccines.

Several studies have suggested that patients with autoimmune conditions may be at increased risk of poor COVID-19 outcomes. There is an urgent need to better clarify the immunogenicity and safety of COVID-19 vaccines in people living with rheumatic disease who use immunomodulatory therapies. Boosters at annual or other frequency are available, and there is a need to understand whether these vaccines can be given concurrently with other routine vaccines.

DETAILED DESCRIPTION:
The COVID-19 pandemic, caused by the coronavirus SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2), has infected a substantial portion of the world population, leading to millions of deaths since its first description in December of 2019. Recently, several SARS-CoV-2 vaccines have shown excellent efficacy and tolerability in the general population and have been either fully approved or given emergency use authorization by the US Food and Drug Administration (FDA), while several other vaccines are in late-stage clinical trials.

Patients with autoimmune conditions, however, particularly those receiving immunomodulatory therapies, have largely been excluded from clinical trials. Yet, certain immunomodulatory therapies have been shown to affect responses to vaccines, with effects varying depending on the medication and type of vaccine. In line with the experience with influenza, pneumococcal and shingles vaccinations in rheumatic disease populations, it is clear that some disease modifying anti-rheumatic drugs (DMARDs) and the immunomodulatory therapies used to treat immune-mediated inflammatory diseases have the capacity to blunt immune responses to COVID-19 vaccines. In addition, a hypothetical concern is that stimulation of the immune system could lead to flares of autoimmune conditions, or new onset autoimmune manifestations. Concerns about flare or disease worsening with vaccination is also substantial among patients themselves, and can sometimes be a reason for vaccine hesitancy or refusal.

Due to recent development and subsequent massive deployment of SARS-CoV-2 vaccines to combat the pandemic, their safety and immunogenicity in patients receiving immunomodulatory therapies had received limited evaluation to date. At the same time, several studies have suggested that patients with autoimmune conditions may be at increased risk of poor COVID-19 outcomes, including hospitalization and death, raising the importance of effective vaccination in this setting. In this context, there is an urgent need to better clarify the immunogenicity and safety of COVID-19 vaccines in people living with rheumatic disease who use immunomodulatory therapies. Additionally, the likelihood that patients will need to be vaccinated in the future again for COVID-19 is high. Boosters at annual or other frequency are likely for all (and have now already been recommended for immunocompromised individuals), and the need to understand whether these vaccines can be given concurrently with other routine vaccines will be important for both patients and clinicians, as well as public health officials. The "vaccine moment" clinically frequently offers the opportunity to give multiple vaccines at one time. Vaccines for other respiratory pathogens (e.g. influenza), hepatitis A, pertussis, and other disease are indicated in large segments of the population, including being of utmost importance in the elderly and those with various chronic conditions and/or immunosuppression. It is imperative to understand whether co-administrated vaccines affect the immunogenicity, efficacy, or safety of COVID-19 vaccines and those vaccines of public health significance given concurrently.

With this background in mind and the momentum of the vaccine campaign in the US to date, whereby the majority of at-risk rheumatology and other populations have received their initial vaccine series, this protocol will focus on evaluating vaccine responses in those receiving a booster mRNA SARS-CoV-2 vaccination. This is important, as boosters are now recommended for all adult patients in the US who have received any prior SARS-CoV-2 vaccination. Further, given a large percentage of rheumatology patients can have sub-optimal or lower immune responses, booster vaccinations will be likely of utmost importance to these and other immunosuppressed groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the inclusion criteria at the time of screening
* Must be 18 years of age or older
* Must live in the United States
* Scheduled for SARS-CoV-2 booster vaccination
* Patients in Rheumatic Disease arm (arm 4) must have inflammatory arthritis (e.g. rheumatoid arthritis, psoriatic arthritis, other) and be receiving stable doses of one of the following medication classes: TNF antagonists, B-cell depletion agents, IL-6 inhibitors, JAK inhibitors, IL-12/23 or IL-23 blockers, IL-17 inhibitors, methotrexate, sulfasalazine, leflunamide, or chronic prednisone (>15mg/day). Stable dosing is defined as no change in dose in the 30 days prior to enrolment.
* For Arms 1-3: patients seen by rheumatologists who do not have active rheumatic disease requiring immunosuppressive therapy. These will include patients with a past history of auto-immune disease that is no longer active, as well as those with other chronic conditions not associated with autoimmune condition such as osteoarthritis, osteoporosis, or other.
* Patients in the Co-administration arms (arms 2 and 3) must meet ACIP recommendations for the use of HAVRIX® (i.e. not previously vaccinated) and BOOSTRIX® (i.e. last immunization >9 years ago).
* Patients who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. completion of the REDCap/diary cards, capable of receiving text messages and/or have a personal email address, return for follow-up visits).

Exclusion Criteria:

* Active infection with SARS-CoV-2 (symptom onset or first positive test in the 14 days prior to recruitment) / disease
* Any known contraindication to SARS-CoV-2 (booster) vaccination, including severe allergy to vaccine components
* Prior use of adenoviral COVID-19 vaccination
* Known or history of HIV/AIDS
* Currently receiving radiation or chemotherapy for any type of malignancy
* Receipt of any immunizations other than SARS-CoV-2 within two weeks prior planned SARS-CoV-2 vaccination, or scheduled within 10 weeks after visit 1
* Significant underlying illness that would be expected to prevent completion of the study (e.g., life-threatening disease likely to limit survival to < 1 year)
* Patients who have a previous history of pericarditis/myocarditis associated with vaccination
* Any other reason that, in the opinion of the site investigator, would interfere with required study related evaluations (e.g. uncontrolled comorbidity)
* Prior receipt of any hepatitis A containing vaccine
* Prior receipt of diphtheria, acellular pertussis, or tetanus vaccination within the last 9 years
* History of physician-diagnosed or laboratory confirmed pertussis within the past 5 years; any history of diphtheria, tetanus disease, or hepatitis A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Ratio of participants' anti-RBD IgG antibodies specific to SARS-CoV-2 measured post-vaccination for those who received only the SARS-CoV-2 booster compared to those who received sequential vaccination with the SARS-CoV-2 booster. | 2 years
  Descriptively evaluate the immunogenicity of anti-spike IgG among patients receiving SARS-CoV-2 booster vaccines alone (Arm 4 N=100) as compared to patients receiving SARS-CoV-2 booster vaccine with sequential vaccination (Arm 1 N=100). The geometric mean concentration ratio (GMC) of Arm 4 to Arm 1 at Week 4 will be reported.
Ratio of participants' anti-RBD IgG antibodies specific to SARS-CoV-2 for those who received sequential vaccination with the SARS-CoV-2 booster compared to those who received a tdap booster co-administered with the SARS-CoV-2 booster. | 2 years
  Descriptively evaluate the immunogenicity of anti-spike IgG among patients receiving SARS-CoV-2 booster vaccines with sequential vaccination (Arm 1 N=100) as compared to patient receiving SARS-CoV-2 booster vaccine with co-administration of BOOSTRIX® (Arm 2 N=100). The geometric mean concentration ratio (GMC) of Arm 1 to Arm 2 at each 4-week interval for Arm 1 (e.g. Week 4, 8, and 36) will be reported.
Ratio of participants' anti-RBD IgG antibodies specific to SARS-CoV-2 for those who received sequential vaccination with the SARS-CoV-2 booster compared to those who received a hepA vaccination co-administered with the SARS-CoV-2 booster. | 2 years
  Descriptively evaluate the immunogenicity of anti-spike IgG among patients receiving SARS-CoV-2 booster vaccines with sequential vaccination (Arm 1 N=100) as compared to patient receiving SARS-CoV-2 booster vaccine with co-administration of HAVRIX® (Arm 3 N=100). The geometric mean concentration ratio (GMC) of Arm 1 to Arm 3 at each 4-week interval for Arm 1 (e.g. Week 4, 8, and 36) will be reported.
Number of participants with solicited localized and general symptoms (Arm 4 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines alone (Arm 4 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine with sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). Number of participants with solicited local and general symptoms that occur within an 8 day period following each vaccine dose administered as assessed by CTCAE will be reported.
Number of participants with unsolicited events (Arm 4 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines alone (Arm 4 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine with sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). Number of participants with unsolicited events occurring within a 31 day period following each vaccine dose administered as assessed by CTCAE will be reported.
Number of medically attended events (Arm 4 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines with either co-administration of BOOSTRIX® (Arm 2 N=100; cell-mediated immunity subset N=50 of first enrolled) or co-administration of HAVRIX® (Arm 3 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). All medically attended events.
Number of confirmed cases of COVID-19 (Arm 4 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines with either co-administration of BOOSTRIX® (Arm 2 N=100; cell-mediated immunity subset N=50 of first enrolled) or co-administration of HAVRIX® (Arm 3 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). Number of confirmed cases of COVID-19 as diagnosed by PCR or antigen-based testing.
Number of potential immune-mediated diseases (Arm 4 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines with either co-administration of BOOSTRIX® (Arm 2 N=100; cell-mediated immunity subset N=50 of first enrolled) or co-administration of HAVRIX® (Arm 3 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). Number of potential immune-mediated diseases (pIMDs; new onset or exacerbation of current).
Number of serious adverse events (Arm 4 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines with either co-administration of BOOSTRIX® (Arm 2 N=100; cell-mediated immunity subset N=50 of first enrolled) or co-administration of HAVRIX® (Arm 3 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). Number of serious adverse events as assessed by CTCAE.
Ratio of participants' anti-RBD IgG antibodies specific to SARS-CoV-2 for those who received a tdap booster co-administered with the SARS-CoV-2 booster compared to those who received sequential vaccination with the SARS-CoV-2 booster. | 2 years
  Descriptively evaluate the immunogenicity of anti-spike IgG among patients receiving SARS-CoV-2 booster vaccine with co-administration of BOOSTRIX® (Arm 2 N=100) as compared to patients receiving SARS-CoV-2 booster vaccine with sequential vaccination (Arm 1 N=100). The geometric mean concentration ratio (GMC) of Arm 2 to Arm 1 at 4 weeks post-vaccination for SARS CoV-2 and BOOSTRIX®.
Ratio of participants' anti-RBD IgG antibodies specific to SARS-CoV-2 for those who received a hepA vaccination co-administered with the SARS-CoV-2 booster compared to those who received sequential vaccination with the SARS-CoV-2 booster. | 2 years
  Descriptively evaluate the immunogenicity of anti-spike IgG among patients receiving SARS-CoV-2 booster vaccine with co-administration of HAVRIX® (Arm 3 N=100) as compared to patients receiving SARS-CoV-2 booster vaccine with sequential vaccination (Arm 1 N=100). The geometric mean concentration ratio (GMC) of Arm 3 to Arm 1 at 4 weeks post-vaccination for dose 2 of HAVRIX® will be reported.
Number of participants with solicited localized and general symptoms (Arm 2 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines with either co-administration of BOOSTRIX® (Arm 2 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). Number of participants with solicited local and general symptoms that occur within an 8 day period following each vaccine dose administered as assessed by CTCAE.
Number of participants with unsolicited events (Arm 2 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines with either co-administration of BOOSTRIX® (Arm 2 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). Number of participants with unsolicited events occurring within a 31 day period following each vaccine dose administered as assessed by CTCAE.
Number of medically attended events (Arm 2 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines with either co-administration of BOOSTRIX® (Arm 2 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). All medically attended events.
Number of confirmed cases of COVID-19 (Arm 2 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines with either co-administration of BOOSTRIX® (Arm 2 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). Number of confirmed cases of COVID-19 as diagnosed by PCR or antigen-based testing.
Number of potential immune-mediated diseases (Arm 2 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines with either co-administration of BOOSTRIX® (Arm 2 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). Number of potential immune-mediated diseases (pIMDs; new onset or exacerbation of current).
Number of serious adverse events (Arm 2 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines with either co-administration of BOOSTRIX® (Arm 2 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). Number of serious adverse events.
Number of participants with solicited localized and general symptoms (Arm 3 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines with either co-administration of HAVRIX® (Arm 3 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). Number of participants with solicited local and general symptoms that occur within an 8 day period following each vaccine dose administered as assessed by CTCAE.
Number of participants with unsolicited events (Arm 3 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines with either co-administration of HAVRIX® (Arm 3 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). Number of participants with unsolicited events occurring within a 31 day period following each vaccine dose administered as assessed by CTCAE
Number of medically attended events (Arm 3 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines with either co-administration of HAVRIX® (Arm 3 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). All medically attended events
Number of confirmed cases of COVID-19 (Arm 3 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines with either co-administration of HAVRIX® (Arm 3 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). Number of confirmed cases of COVID-19 as diagnosed by PCR or antigen-based testing
Number of potential immune-mediated diseases (Arm 3 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines with either co-administration of HAVRIX® (Arm 3 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). Number of potential immune-mediated diseases (pIMDs; new onset or exacerbation of current).
Number of serious adverse events (Arm 3 to Arm 1) | 2 years
  Descriptively evaluate the safety and reactogenicity of patients receiving SARS-CoV-2 booster vaccines with either co-administration of HAVRIX® (Arm 3 N=100; cell-mediated immunity subset N=50 of first enrolled) as compared to patients receiving SARS-CoV-2 booster vaccine sequential vaccination (Arm 1 N=100; cell-mediated immunity subset N=50 of first enrolled). Number of serious adverse events as assessed by CTCAE.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Center for Rheumatic Diseases, Northport, Alabama
  - Sun Valley Arthritis, Peoria, Arizona
  - Ocean Wellness Center, Miami Gardens, Florida
  - Southwest Florida Rheumatology, Riverview, Florida
  - St. Luke's Rheumatology, Boise, Idaho
  - Ravenswood Rheumatology, Chicago, Illinois
  - University Medical Center - New Orleans/LSU, New Orleans, Louisiana
  - St. Paul Rheumatology, Eagan, Minnesota
  - Jayashree Sinha, MD, Clovis, New Mexico
  - Oregon Health & Science University, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Cumberland Rheumatology, Crossville, Tennessee
  - Advanced Rheumatology of Houston, Woodland, Texas

IPD SHARING:
Plan to Share IPD: Undecided